CLINICAL TRIAL: NCT06342804
Title: An Open-label Crossover Study With 2 Treatments (Fasting and Fed Conditions), 2 Periods, 2 Sequences to Evaluate the Effect of Food Intake on the Bioavailability of 4-MUST, Tablets, 128 mg at a Single Dose of 256 mg in Healthy Volunteers
Brief Title: Food Effect on the Bioavailability of 4-MUST, Tablets, 128 mg
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Valenta Pharm JSC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: GIB-01-02-2023
Record Dates: First submitted 2024-03-11; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-02

CONDITIONS: Cholecystitis
MeSH Terms: conditions — Cholecystitis | interventions — Postprandial Period

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AB sequence (Experimental): Group 1 (sequence AB) will take the drug on an empty stomach in Period I and after a meal in Period II
  Interventions: Drug: 4-MUST, 2 tablets, fasted; Drug: 4-MUST, 2 tablets, after meals
- BA sequence (Experimental): Group 2 (BA sequence) will take the drug after a meal in Period I and on an empty stomach in Period II
  Interventions: Drug: 4-MUST, 2 tablets, fasted; Drug: 4-MUST, 2 tablets, after meals

INTERVENTIONS:
Drug: 4-MUST, 2 tablets, fasted — 2 tablets (256 mg), fasted
  Other Names: 4-methylumbelliferyl trimebutine sulfate
Drug: 4-MUST, 2 tablets, after meals — 2 tablets (256 mg), after meals
  Other Names: 4-methylumbelliferyl trimebutine sulfate

SUMMARY:
Primary objective of the study: evaluation of the effect of food intake on the bioavailability of 4-MUST, tablets, 128 mg (Valenta Pharm JSC) after a single oral administration on an empty stomach and after a meal, at a dose of 256 mg (two tablets).

Additional aim of the study: evaluation of pharmacokinetic parameters, safety and tolerability of 4-MUST, tablets, 128 mg (Valenta Pharm JSC) in healthy volunteers after a single oral administration on an empty stomach and after a meal, at a dose of 256 mg (two tablets).

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary and handwritten informed consent form signed by a healthy volunteer to participate in the study prior to any of the study procedures;
2. Males and females between the ages of 18 and 45 years (inclusive) of Caucasian race;
3. Verified diagnosis of "healthy" (absence of abnormalities according to the data of clinical, laboratory, instrumental methods of examination stipulated by the protocol);
4. Blood pressure (BP) level: systolic blood pressure (SBP) from 99 to 129 mmHg (inclusive), diastolic blood pressure (DBP) from 70 to 89 mmHg (inclusive);
5. Heart rate (HR) from 60 to 89 beats/min (inclusive);
6. Respiratory rate (RR) from 12 to 20 per 1 minute (inclusive);
7. Body temperature from 36.0°C to 36.9°C (inclusive);
8. Body mass index (BMI) of 18.5 kg/m2 ≤ BMI ≤ 30 kg/m2, with body weight ≥ 55 kg for males and ≥ 45 kg for females;
9. Agreement to use adequate contraceptive methods throughout the study and for 30 days after completion of the study, for women of preserved reproductive potential, a negative urine pregnancy test result.

Noninclusion Criteria:

1. Aggravated allergic history;
2. Hypersensitivity to gimecromone and trimebutine and/or excipients included in the investigational medicinal product in anamnesis;
3. Drug intolerance to hymecromone and trimebutine and/or excipients included in the investigational medicinal product in the anamnesis;
4. Hereditary galactose intolerance, lactase deficiency or glucose-galactose malabsorption in the anamnesis;
5. Chronic diseases of the kidney, liver, gastrointestinal tract (GIT), cardiovascular, lymphatic, respiratory, nervous, endocrine, musculoskeletal, genitourinary and immune systems, as well as skin, hematopoietic and visual organs;
6. A history of GI surgery (except for appendectomy at least 1 year prior to screening);
7. Diseases/conditions that, in the opinion of the investigator, may affect the absorption, distribution, metabolism, or excretion of the investigational drug;
8. Acute infectious diseases less than 4 weeks prior to screening;
9. Intake of drugs that have a significant effect on hemodynamics and drugs that affect liver function (barbiturates, omeprazole, cimetidine, etc.) less than 2 months before screening;
10. Regular intake of a medicine less than 2 weeks prior to screening and single intake of a medicine less than 7 days prior to screening (including over-the-counter medicines, vitamins, supplements, herbs);
11. Blood or plasma donation less than 3 months prior to screening;
12. Use of hormonal contraceptives (in women) less than 2 months prior to screening;
13. Use of depot injections of any medicine less than 3 months prior to screening;
14. Pregnancy or lactation period; positive urine pregnancy test for women of preserved reproductive potential;
15. Women of preserved reproductive potential with a history of unprotected sexual intercourse within 30 days prior to study medication with an unsterilized partner;
16. Participation in another clinical trial less than 3 months prior to screening or concurrent with the present study;
17. Intake of more than 10 units of alcohol (1 unit of alcohol is equivalent to 500 mL of beer, 200 mL of wine, or 50 mL of spirits) per week in the last month prior to inclusion in the study or history of alcoholism, drug abuse, or medicine abuse;
18. Smoking more than 10 cigarettes per day currently, or a history of smoking the indicated number of cigarettes in the 6 months preceding screening; failure to agree to abstain from smoking for the duration of the hospital stay;
19. Consumption of alcohol, caffeine, and xanthine-containing products in the 7 days prior to taking the study drug;
20. Consumption of citrus fruits, cranberries, rose hips and products containing them, preparations or products containing St. John's wort - 7 days before taking the study drug;
21. Dehydration due to diarrhea, vomiting, or other cause within the last 24 hours prior to taking the study drug;
22. Positive blood test result for antibodies to human immunodeficiency virus (HIV) 1 and 2, antibodies to Treponema pallidum antigens, hepatitis B surface antigen (HBsAg), antibodies to hepatitis C virus antigens at screening;
23. Positive result of rapid test for coronavirus disease pathogen 2019 (Coronavirus disease 2019, COVID-19) at screening;
24. Clinically significant electrocardiogram (ECG) abnormalities with a history and/or at screening;
25. Positive urinalysis for narcotics and potent drugs at screening;
26. Positive breath alcohol vapor test at screening;
27. Scheduling a hospital stay during the study period, for any reason other than hospitalization required by this protocol;
28. Failure or inability to comply with protocol requirements, follow protocol procedures, diet and activity regimen.
29. Vulnerable group of volunteers: medical, pharmacy and dental students, clinical and laboratory assistants, pharmaceutical company employees, military personnel and prisoners, care home residents, low-income and unemployed, minorities, homeless, vagrants, refugees, persons in foster care, persons unable to consent, and law enforcement officers;
30. Other conditions that, in the opinion of the Investigator, would preclude the inclusion of the volunteer in the study or could result in early withdrawal of the volunteer from the study, including fasting or a special diet (e.g., vegetarian, vegan, limited table salt) or a special lifestyle (night work, extreme physical exertion).

Exclusion criteria:

1. The volunteer refuses to participate in the study;
2. Failure of the volunteer to comply with the rules of participation in the study (skipping study procedures, independent use of drugs prohibited in the study, violation of dietary and lifestyle restrictions, etc.);
3. Causes/occurrence of situations during the study that jeopardize the safety of the volunteer (e.g. hypersensitivity reactions, etc.);
4. Volunteers selected for participation in the study in violation of the inclusion/non-inclusion criteria;
5. Development of severe adverse event and/or a serious adverse event in a volunteer during the course of the study;
6. Volunteer is receiving or requires treatment that may affect the pharmacokinetic parameters of the study drug;
7. Missing collection of 2 or more consecutive blood samples or 3 x or more blood samples during the same Study Period;
8. Occurrence of vomiting/diarrhea within 6 h after administration of study drug;
9. Positive urine test for narcotics and potent drugs;
10. Positive breath alcohol vapor test;
11. A positive pregnancy test in women;
12. Positive test for COVID-19;
13. Occurrence of other reasons during the study that prevent the conduct of the study according to the protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics - Cmax | From 0 to 48 hours (days 1-3 and 8-10)
  Maximum plasma concentration (Cmax) of N-desmethyltrimebutin, 4-methylumbelliferone sulfate and 4-methylumbelliferone
Pharmacokinetics - tmax | From 0 to 48 hours (days 1-3 and 8-10)
  Time to reach Cmax (tmax) of N-desmethyltrimebutin, 4-methylumbelliferone sulfate and 4-methylumbelliferone
Pharmacokinetics - AUC0-t | From 0 to 48 hours (days 1-3 and 8-10)
  Area under the plasma concentration-time curve from time 0 to t (AUC0-t) of N-desmethyltrimebutin, 4-methylumbelliferone sulfate and 4-methylumbelliferone
Pharmacokinetics - AUC0-inf | From 0 to 48 hours (days 1-3 and 8-10)
  Area under the plasma concentration-time curve from time 0 to infinity (AUC0-inf) of N-desmethyltrimebutin, 4-methylumbelliferone sulfate and 4-methylumbelliferone
Pharmacokinetics - AUC ratio | From 0 to 48 hours (days 1-3 and 8-10)
  The ratio of the area under the concentration-time curve over the observation time to the calculated area under the concentration-time curve from zero to infinity
Pharmacokinetics - t1/2 | From 0 to 48 hours (days 1-3 and 8-10)
  Elimination half-life (t1/2) of N-desmethyltrimebutin, 4-methylumbelliferone sulfate and 4-methylumbelliferone
Pharmacokinetics - kel | From 0 to 48 hours (days 1-3 and 8-10)
  Elimination constant (kel) of N-desmethyltrimebutin, 4-methylumbelliferone sulfate and 4-methylumbelliferone
Pharmacokinetics - MRT | From 0 to 48 hours (days 1-3 and 8-10)
  Mean residence time (MRT) of N-desmethyltrimebutin, 4-methylumbelliferone sulfate and 4-methylumbelliferone
Pharmacokinetics - Vd | From 0 to 48 hours (days 1-3 and 8-10)
  Volume of distribution of N-desmethyltrimebutin, 4-methylumbelliferone sulfate and 4-methylumbelliferone
Pharmacokinetics - Cmax/AUC0-t | From 0 to 48 hours (days 1-3 and 8-10)
  The ratio of the maximum concentration to the area under the concentration-time curve during the observation period
Pharmacokinetics - f' | From 0 to 48 hours (days 1-3 and 8-10)
  f' - relative bioavailability (AUC(0-t)(fed)/AUC(0- t)(fasting))
Pharmacokinetics - f'' | From 0 to 48 hours (days 1-3 and 8-10)
  f'' is the relative absorption rate (Cmax(fed)/Cmax(fasting))
Bioavailability - ratio of Cmax | From 0 to 48 hours (days 1-3 and 8-10)
  Ratio of geometric mean Cmax for N-desmethyltrimebutin, 4-methylumbelliferone sulfate and 4-methylumbelliferone in fasted and fed conditions (with 90% confidence intervals)
Bioavailability - ratio of AUC0-t | From 0 to 48 hours (days 1-3 and 8-10)
  Ratio of geometric mean AUC0-t for N-desmethyltrimebutin, 4-methylumbelliferone sulfate and 4-methylumbelliferone in fasted and fed conditions (with 90% confidence intervals)
Bioavailability - ratio of AUC0-inf | From 0 to 48 hours (days 1-3 and 8-10)
  Ratio of geometric mean AUC0-inf for N-desmethyltrimebutin, 4-methylumbelliferone sulfate and 4-methylumbelliferone in fasted and fed conditions (with 90% confidence intervals)

SECONDARY OUTCOMES:
Adverse event type | From day -14 - day -1 (screening) to day 16 ± 1 (end of the study)
  Adverse events will be assessed by complaints, results of physical examination, results of heart rate and blood pressure assessment, results of respiratory rate assessment, body temperature, laboratory monitoring (clinical blood count, biochemical blood count, urinalysis), electrocardiography; adverse events will be classified in accordance to MedDRA.
Adverse event frequency | From day -14 - day -1 (screening) to day 16 ± 1 (end of the study)
  Number and frequency of adverse events registered during the study
Adverse event severety | From day -14 - day -1 (screening) to day 16 ± 1 (end of the study)
  Severity of adverse events registered during the study
Drop-outs associated with adverse events | From day -14 - day -1 (screening) to day 16 ± 1 (end of the study)
  The number of cases of early termination of participation in the study due to the development of adverse events and/or serious adverse events associated with the study drug

CONTACTS AND LOCATIONS:
Locations (1):
- Federal Budgetary Institution of Science "North-Western Scientific Center for Hygiene and Public Health", Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No